CLINICAL TRIAL: NCT05185635
Title: Validating Neuropsychological Tests Among Healthy Spanish-Speaking Adults: A Pilot Study
Brief Title: Validating Neuropsych Tests in Spanish-speakers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rehabilitation Hospital of Indiana (Other)
Responsible Party: Principal Investigator, Patricia Garcia, Neuropsychologist, Rehabilitation Hospital of Indiana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 11390
Record Dates: First submitted 2021-09-29; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Neuropsychology; Testing
Keywords: Spanish-speakers

STUDY DESIGN:
Intervention Model Description: This project is an initial cross-sectional study of 40 Spanish-speaking subjects to generate pilot normative neuropsychological performance data that will be used in the future in grant submissions and as an initial feasibility platform for larger scale research projects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Spanish-speakers (Experimental)
  Interventions: Diagnostic Test: Neuropsychological testing

INTERVENTIONS:
Diagnostic Test: Neuropsychological testing — potential participants will complete the following: Mini-Mental State Examination (MMSE), Patient Health Questionnaire-9 (PHQ-9) and Generalized Anxiety Disorder 7- item (GAD-7) as part of the screening process. Additionally to the pre-screening instruments, participants will complete the following neuropsychological tests: Bi-dimensional Acculturation Scale, Bilingual Dominance Scale, Verbal Fluency Tests, Boston Naming Test, Symbol Digit Modalities Test, Brief Test of Attention, Who-UCLA Auditory Verbal Learning Test, Rey-Osterrieth Complex Figure, Modified Wisconsin Card Sorting Test, Stroop Color and Word Test, Trail Making Test, Word Accentuation Test, Clock Drawing Task, Bells Test, Test of Memory Malingering, and the Five Point Test.

SUMMARY:
The proposed pilot further emphasizes the need for collecting language and demographic specific norms for Spanish-speaking Latino individuals in the U.S. by developing new normative test data for this demographic population. The study looks to contribute to minimize healthcare disparities and inaccurate test interpretations, which can have direct implications on diagnosis and treatment. This study will allow us to develop new neuropsychological test norms for predominantly Spanish-speaking adults by establishing expected cognitive performance on a battery of frequently used neuropsychological tests. As such, the current study will help fill a large gap in the literature pertaining to neuropsychological assessment of Spanish-Speakers living in the U.S., as well as produce data of clinical utility for providers working with this population. Finally, this pilot could serve as a model to eventually extend it to other non-English speaking populations in the US.

DETAILED DESCRIPTION:
Hispanics/Latinos are now recognized as the largest and fastest growing ethnic/racial minority group in the United States (U.S.). By 2017, the Hispanic/Latino population reached nearly 60 million comprising 18% of the total U.S. population. Current projections indicate that Hispanic/Latinos will reach almost 111 million, making up 28% of the total U.S. population by 2060.

Clinical neuropsychologists must be equipped with the right tools to accurately serve the rapidly growing Hispanic/Latino population in the US. Findings from normative data studies in foreign countries emphasize the need for developing language and demographic specific norms for Spanish-speaking Hispanics in the US. This is particularly relevant given recent literature indicating that factors such as ethnicity, language, quality of education, degree of acculturation, and bilingualism can have a profound impact on neuropsychological test performance. Within participants that self-identify as primarily Spanish-speaking, language performance has been positively associated with greater Spanish vs. English language dominance and completing education outside the U.S., whereas other cognitive abilities have a negative association with the same variables.

The proposed pilot further emphasizes the need for collecting language and demographic specific norms for Spanish-speaking Latino individuals in the U.S. by developing new normative test data for this demographic population. The study looks to contribute to minimize healthcare disparities and inaccurate test interpretations, which can have direct implications on diagnosis and treatment. This study will allow us to develop new neuropsychological test norms for predominantly Spanish-speaking adults by establishing expected cognitive performance on a battery of frequently used neuropsychological tests. As such, the current study will help fill a large gap in the literature pertaining to neuropsychological assessment of Spanish-Speakers living in the U.S., as well as produce data of clinical utility for providers working with this population. Finally, this pilot could serve as a model to eventually extend it to other non-English speaking populations in the US.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 to 80 years of age
* Have been living in the US for at least 1 year (12 continuous months)
* Identify Spanish as their primary and/or dominant language
* Have at least one year of formal education
* Be able to read and write at the time of evaluation in Spanish
* a score of ≥23 on the Mini-Mental State Examination (MMSE)
* score of ≤10 on the Patient Health Questionnaire-9 (PHQ-9)
* score of ≤10 on the generalized anxiety disorder (GAD-7)

Exclusion Criteria:

* History of neurodevelopmental disorder
* History of learning disorder
* Past or present neurologic condition
* Past or present chronic medical condition that may affect cognition (i.e. metabolic syndrome, chronic heart failure, sleep apnea)
* Past or present use of psychotropic medications that may affect cognition
* Past or present history of substance abuse or dependence
* Past or present history of psychiatric disorder
* Presence of severe sensory deficits, such as loss of hearing or vision

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE) | Up to 5 months
  The Mini-Mental State Examination (MMSE) is well known cognitive screening tool that is widely used in neuropsychological clinical practice. Several reports have used this rapid test as a baseline measure to obtain reliable diagnoses when cognitive impairment is suspected. The MMSE has many benefits, particularly its rapid application and high sensitivity and specificity in relation to cognitive dysfunction.
Patient Health Questionnaire (PHQ-9) | Up to 5 months
  The Patient Health Questionnaire is a self-administered assessment tool used to screen specifically for the presence depression.
Generalized Anxiety Disorder(GAD-7) | Up to 5 months
  The Generalized Anxiety Disorder 7-item test is a useful self-report measure with strong criterion validity for identifying probable cases of GAD.
Bidimensional Acculturation Scale (BAS) | Up to 5 months
  The Bidimensional Acculturation Scale is a 24-item measure that assesses an individual's level of acculturation to Hispanic culture and to non-Hispanic culture.
Gradient Bilingual Dominance Scale | Up to 5 months
  The Bilingual Dominance Scale (BDS; Dunn & Tree, 2009) is a 12 item self-report measure that can be used to quantify the language dominance of bilingual participants.
Verbal Fluency Tests | Up to 5 months
  Verbal fluency tests (VFT) are commonly used measures both in clinical practice and research due to their sensitivity to brain damage. There are multiple variations of the VFT, but the two more commonly used paradigms measure letter and semantic fluency. In the letter VFT, participants are asked to produce as many words as possible that begin with a certain letter within a 60 second time limit. In the semantic VFT, participants are required to produce as many words as s/he can that belong to a category within the same 60 second timeframe.
Standard Form of the Boston Naming Test | Up to 5 months
  The Boston Naming Test requires examinees to denominate 60 pictures, which are presented in order of increasing difficulty. If the participant does not spontaneously provide the correct response, the examiner provides a prompt in the form of a semantic cue or phonological cue
The Symbol Digit Modalities Test | Up to 5 months
  The Symbol Digit Modalities Test is a timed measure that requires participants to convert symbols (shaped geometric figures) into numbers, as quickly as possible.
Brief Test of Attention | Up to 5 months
  The Brief Test of Attention test consists of two equivalent forms that are administered consecutively (Forms N and L). In the N form, the subject hears a list of 10 series of letters and numbers that are intercalated, after which the subject must indicate how many numbers were mentioned. Subsequently, in the form L, the subjects are presented the same list series, but this time the subject must indicate how many letters were mentioned.
WHO-UCLA Auditory Verbal Learning Test (WHO-UCLA AVLT) | Up to 5 months
  The WHO-UCLA Auditory Verbal Learning Test (AVLT) is a measure of verbal learning and memory that consists of 15 words selected from a standardized lexicon of 250 universally familiar concepts . The 15-item word list is repeated across five learning trials, and patients are to complete immediate recall, do an interference task, a short-delay free-recall, a 20-min delay, and then another free recall, followed by forced choice.
Rey-Osterrieth Complex Figure | Up to 5 months
  The Rey-Osterrieth Complex Figure Test is a measure of visual perception, visual-spatial constructional ability, and visual memory that was developed by Swiss psychologist Andre Rey in 1941. For the purpose of the present study, the Spanish-language ROCF manual scoring guidelines will be followed (Rey, 2009).
Modified Wisconsin Card Sorting Test (M-WCST) | Up to 5 months
  The Modified Wisconsin Card Sorting Test consists of four stimulus cards and 48 response cards. Each card varies in shape (cross, circle, triangle or star), color (red, blue, yellow or green), and number (one to four). The first participant's response is always considered right, and during the administration, the examiner informs him/her whether their response is correct or incorrect until the participant accurately classifies six consecutive cards in each category. Then, the examiner indicates that the rules have changed and to try to "find another rule." If the second category chosen differs from what was chosen in the first, it is considered correct. The test continues until all six categories are classified or until having used the whole card deck
Stroop Color-Word Interference Test | Up to 5 months
  The Stroop Color and Word test consists of three pages, each with 100 components randomly organized into five columns. The subject has 45 seconds to read aloud, as quickly as possible, the columns from left to right. The sheet on words is formed by the words "Red," "Green," and "Blue" in black ink, and the score is the number of words read correctly. For the sheet containing only colors, there are groups of four X's ("XXXX") printed in blue, green, and red. The score is the number of elements properly named. Finally, the last list consists of the three words of the first printed page in the colors of the second, with words being incongruent with the color of the ink. The task is to name the ink color, inhibiting the reading of the word, and the score is the number of correctly named elements.
Trail Making Test | Up to 5 months
  The Trail Making Test is a times measure consists of two parts: TMT-A and B. In the TMT-A the participant must draw a line, as quickly as they can, connecting 25 numbers in ascending order, which are circled and randomly distributed on a sheet of paper. The task requirements are similar for the TMT-B, except that the person alternates between numbers and letters the latter being significantly more difficult
Word Accentuation Test-Chicago (WAT-C) | Up to 5 months
  The Word Accentuation Test is a reading test utilized to estimate premorbid cognitive ability among Spanish-speaking individual's ages 29-73 years.
Clock Drawing Test | Up to 5 months
  The Clock Drawing Test is a measure that screens for dementia as well as for visuospatial, constructional, and visual planning difficulties. T
Bells Test | Up to 5 months
  The Bells Test is used to detect visual inattention in children and adults and it consists of a 21.5 × 28 cm sheet of paper on which seven lines of 35 distractor figures (e.g., bird, key, apple, mushroom, car) and five target figures (bells) are presented.
Test of Memory Malingering (TOMM II) | Up to 5 months
  The Test of Memory Malingering is a visual recognition test designed to help distinguish between bona fide and malingered memory impairments.
Five Point Test | Up to 5 months
  The Five Point Test is a measure that requires production of novel designs under time constraints. Patients are asked to produce as many different figures as possible by connecting the dots within each rectangle.

IPD SHARING:
Plan to Share IPD: No